CLINICAL TRIAL: NCT03582293
Title: Tranexamic Acid to Prevent OpeRation in Chronic Subdural Hematoma. A Double-blind, Placebo-controlled, Multicentre, Randomized Controlled Clinical Trial
Brief Title: Tranexamic Acid to Prevent OpeRation in Chronic Subdural Hematoma
Acronym: TORCH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Prof. dr. W.Peter Vandertop, chair Neurosurgery, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL63794.018.18
Record Dates: First submitted 2018-06-19; First posted 2018-07-11 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Hematoma, Subdural, Chronic
Keywords: Tranexamic Acid; Antifibrinolytic Agents
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Tranexamic Acid; Tablets

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, multicentre, randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid (Active Comparator): Tranexamic acid 500mg two times a day orally for a total of 28 days
  Interventions: Drug: Tranexamic Acid 500Mg Tablet
- PLACEBO (Placebo Comparator): Placebo capsules two times a day orally for a total of 28 days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Tranexamic Acid 500Mg Tablet — orally twice daily for 28 days
  Other Names: Cyklokapron
  Arms: Tranexamic Acid
Drug: Placebo oral capsule — Oral placebo capsule two times a day for a total of 28 days
  Arms: PLACEBO

SUMMARY:
Rationale: Chronic subdural hematoma (cSDH) is a frequently occurring disease, occurring mainly in the elderly. Surgical evacuation is effective, but also associated with life-threatening risks. In these old, often frail, patients with multi-comorbidity, surgery also comes with significant risks for future cognitive functioning and therefore, loss of independency. In five small retrospective series, tranexamic acid (TXA), an antifibrinolytic drug, showed a beneficial effect on the spontaneous resolution of the hematoma and, with that, the necessity for surgery. This randomised, placebo-controlled clinical trial aims to prove the efficacy of TXA.

Objectives: Primarily to evaluate the efficacy of TXA to prevent surgery for cSDH. Secondarily to evaluate the efficacy of TXA to reduce cSDH volume, neurological impairment (mNIHSS), the incidence of falling incidents, the mortality rate, the use of care and health-related costs (iMCQ and iPCQ), to improve cognitive functioning (MOCA), performance in activities of daily living (Barthel and Lawton-Brody), functional outcome (mRS), the level of quality of life.

Study design: Double-blind placebo-controlled multicentre randomized clinical trial.

Study population: All patients, age 50 and above, diagnosed with cSDH for whom a conservative treatment is selected as primary treatment strategy.

Intervention: The intervention group will receive oral TXA 500mg twice daily for 4 weeks, the control group will receive a placebo twice daily. The TXA or placebo treatment is additional to standard care.

Main study endpoint: The number of patients requiring surgery within 12 weeks after start treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients will use the study medication twice daily for four weeks. Follow-up is at 4, 8and 12 weeks with a standard CT-scan of the head, outpatient clinic visits and 4 patient-reported questionnaires. These outpatient clinic visits are standard care; the third CT-scan, the questionnaires and extra clinical tests are extra. Each patient may benefit from the study if the study medication proves effective in preventing surgery for cSDH, whereas the risk of potential side effects of the medication is slight (e.g. the risk of thromboembolic events is only 0.01-0.1%). Surgery remains a possibility for those patients in whom study medication is not effective.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE Chronic subdural hematoma (cSDH) is a frequently occurring neurological disease of the elderly and common in daily neurosurgical practice. It consists of an extracerebral encapsulated collection of mostly liquefied old hematoma, located between the dura and arachnoid. The original small, and often asymptomatic, haemorrhage is caused by rupture of a bridging vein after, often minor, head trauma. Due to generalized cerebral atrophy, increased venous fragility, and the more frequent use of anticoagulation therapy, older people are more at risk of developing a cSDH.

During several weeks, the original hematoma is encapsulated by a membrane consisting of weak neocapillaries from where recurrent small bleedings occur. The pathophysiological mechanism is thought to be a problem in the local haemostasis due to fibrin degradation products of the original small hematoma that inhibit further haemostasis in the subdural space. Together with an osmotic draw of water, owing to its high protein content, this results in growth of the hematoma. Therefore, it usually takes several weeks for the cSDH to grow and become symptomatic.

Signs and symptoms arise due to compression of brain tissue. These can be generalised, such as headaches, light-headedness, cognitive disturbances, apathy, somnolence, seizures, frequent falling and depression. Also focal deficits, such as dysphasia, motor weakness or sensory disturbances, can be symptoms of a cSDH.

The current incidence of cSDH is estimated to be 15/100,000 per year. The number of patients with cSDH is expected to increase considerably in the near future due to the continuing growth of the elderly population, and the increase in the use of anticoagulation and anti-aggregation therapy. By 2030, the incidence is expected to rise up to 20/100,000 per year, thus making cSDH the most common neurosurgical condition in adults. In The Netherlands, this comes down to 3,600 new patients each year.

Treatment Treatment options are conservative and surgical. Conservative treatment currently consists of a wait-and-scan policy in which the patient is regularly monitored for neurological deterioration and growth of the hematoma on follow-up imaging. Anticoagulation and antiplatelet therapy is discontinued in low-risk patients, based on individual risk-benefit assessment and the discretion of the treating physician. If the clinical condition of the patient worsens, the indication for surgical evacuation of the hematoma is re-evaluated.

Spontaneous resolution of cSDH with a conservative treatment occurs in approximately 2.5% of patients, and is therefore relatively rare. Of all patients diagnosed with cSDH in The Netherlands, about 50% is primarily treated conservatively. Of these, around 75% still need an operation (own data). If the symptoms are serious or worsen over time, surgical evacuation of the hematoma is currently the designated therapy. This therapy is an effective treatment, but is also associated with life-threatening risks. In these old, often frail, patients with multi-comorbidity, surgery comes with significant risks for future cognitive functioning and, therefore, loss of independency. In a large series of 1205 patients, symptomatic recurrence after surgery was 9%, mortality 2% and unfavourable functional outcome 22%.

Outcome measurement Studies evaluating quality of life and functional outcome with cSDH patients are scarce. The modified Rankin Scale (mRS) score is usually the only clinical outcome parameter. A literature search for quality of life in cSDH results in only two clinical studies. The first used the postoperative mRS, Barthel Index and Sickness Impact Profile as outcome measurements; the second used a pre- and postoperative Karnofsky Performance Score.

Tranexamic acid As hyperfibrinolysis is thought to play a role in the liquefaction and enlargement of cSDH, pharmaceutical options to block fibrinolysis have been explored in an effort to eliminate the necessity for surgery. The use of tranexamic acid (TXA), an antifibrinolytic drug, has so far been reported in five small series. In the first retrospective series, a total of 21 patients were treated with TXA, of whom three after primary burr hole surgery. In none of these 21 patients, additional surgery was necessary. The second, a prospective pilot study in 14 patients, showed a 41% reduction of cSDH after surgery, and an additional 91% residual volume reduction on CT after 90 days, during oral TXA treatment of 650 mg per day, for a mean (SD) duration of 90 (27) days, without recurrence, re-expansion, or any complicating venous thromboembolisms. The third study, a case report series of three patients treated with 650mg TXA per day for one month after surgery for cSDH, showed no recurrences and thromboembolic complications. The fourth, a case report of one patient successfully treated primarily with TXA, was recently published, and finally, in the abstract of a Asian article, the authors conclude that administration of Gorei-San, a Japanese herbal Kampo medicine, combined with TXA has the potential to prevent recurrences of cSDH.

With these limited, however promising, data no definitive conclusion can be made regarding the role of TXA in the treatment of cSDH. Therefore, a prospective study evaluating the efficacy and safety of TXA is needed. Currently, two prospective trials (the TRACS study and the TRACE study are running in an effort to answer this question. The first study, a phase 2b trial with the aim to provide preliminary data required to plan a larger phase III trial, excludes patients using anticoagulants. These patients comprise a significant portion of the cSDH patient population, and therefore, the results of the TRACS study will be difficult to extrapolate to the future care of all cSDH patients. The second study (TRACE) is a randomised, observer blinded trial, investigating the value of treating cSDH patients with TXA after surgery. This is a different patient population than proposed in the investigators' trial, in which they plan to include only patients in whom the primary treatment is conservative. Also, both trials are set up with a primary radiological outcome parameter and therefore potentially provide insufficient clinically relevant information.

This phase III trial aims to investigate the efficacy and safety of TXA as an addition to a primary conservative treatment of cSDH, in an effort to prevent surgery for cSDH. Since surgical treatment under general anaesthesia and a hospital admittance of a minimum of two days is associated with significant morbidity, as described earlier, the investigators assume that preventing surgery also prevents deterioration of patients' quality of life. This trial is also the first in describing functional outcome and quality of life of cSDH patients in a prospective manner. Since the target population partially comprises patients with a depressed level of consciousness, and patients using anticoagulants and antiplatelets, these patient groups will be included in this trial as well.

ELIGIBILITY:
Inclusion Criteria:

* On CT confirmed cSDH
* Primary conservative treatment, based on clinical symptoms: Glasgow Coma Scale score >=14, mNIHSS score <=4 and a stable neurological deficit (no new, or progression of, symptoms between the assessment by the neurologist and the assessment by the neurosurgeon).

Exclusion Criteria:

Primary surgical treatment based on one or more of the following symptoms or parameters: medically intractable headache, midline shift >10mm, imminent death within 24 hours;

* Structural causes for subdural haemorrhage, e.g. arachnoid cysts, cortical vascular malformations and a history of cranial surgery <1year;
* Aneurysmal subarachnoid haemorrhage;
* Active treatment for deep vein thrombosis, pulmonary embolism or cerebral thrombosis (secondary prophylaxis is not considered to be active treatment);
* Active intravascular clotting or disseminated intravascular coagulation;
* Known hypersensitivity or allergy to TXA or to any of the ingredients;
* History of a blood coagulation disorder (hypercoagulability disorder);
* History of severe impairment of renal function (eGFR <30ml/min or serum creatinine >150μmol/L);
* History of anaemia (haemoglobin <6mmol/L);
* History of convulsions;
* History of inability to safely swallow oral medication.
* Inability to obtain informed consent from the patient or legal representative (when the patient has a depressed level of consciousness as described in paragraph 11.2), including language barrier;

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Estimated)
Dates: Start 2018-06-19 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
surgery for cSDH | within 12 weeks after start of treatment
  number of patients who need to undergo surgery for cSDH

SECONDARY OUTCOMES:
cSDH volume | at four, eight and 12 weeks
  change in cSDH volume (in ml) on follow-up CT scan of the head
neurological impairment | at four, eight and 12 weeks
  neurological impairment measured with the modified National Institutes of Health Stroke Scale (mNIHSS) score, range 0 (normal) to 31 (severe neurological deficit)
falling incidents | during the 12 week study period
  number of falling incidents during study period
cognitive functioning | at four, eight and 12 weeks
  cognitive functioning measured with the Montreal Cognitive Assessment (MOCA) test, range 0 - 30, with a score of 26 and higher generally considered normal.
performance in activities of daily living 1 | at 12 weeks
  performance in activities of daily measured with the Barthel Index scale (range 0-20, with lower scores indicating increased disability)
functional outcome | at 12 weeks
  functional outcome measured with the modified Rankin Scale (mRS) score, range 0 (no symptoms) to 6 (death)
patient health status 1 | at 12 weeks
  quality of life measured with the patient-reported Short Form Health Survey questionnaire (SF-36; eight scaled scores, range 0 (maximum disability) -100 (no disability).
mortality rate | at 12 weeks
  number and percentage of deaths during study period
use of care | during the 12 week study period
  use of care measured with the Medical Consumption Questionnaire (iMCQ), which includes questions related to frequently occurring contacts with health care providers
performance in activities of daily living 2 | at 12 weeks
  performance in activities of daily measured with the Lawton-Brody scale, range 0 (low function, dependent) to 8 (high function, independent).
health-related costs | during the 12 week study period
  health-related costs measured with the Productivity Cost Questionnaire (iPCQ), a standardized instrument including three modules for measuring and valuing productivity losses of paid work due to 1) absenteeism and 2) presenteeism and productivity losses related to 3) unpaid work.
patient health status 2 | at 12 weeks
  quality of life measured with the five dimensional EuroQol questionnaire (EQ-5D-3L, five dimensions with each 3 levels: 1-no problems, 2-some problems, and 3-extreme problems).

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sambasivan M. An overview of chronic subdural hematoma: experience with 2300 cases. Surg Neurol. 1997 May;47(5):418-22. doi: 10.1016/s0090-3019(97)00188-2. PMID 9131021
- [Background] Tagle P, Mery F, Torrealba G, Del Villar S, Carmona H, Campos M, Mendez J, Chicharro A. [Chronic subdural hematoma: a disease of elderly people]. Rev Med Chil. 2003 Feb;131(2):177-82. Spanish. PMID 12708256
- [Background] Adhiyaman V, Asghar M, Ganeshram KN, Bhowmick BK. Chronic subdural haematoma in the elderly. Postgrad Med J. 2002 Feb;78(916):71-5. doi: 10.1136/pmj.78.916.71. PMID 11807186
- [Background] Balser D, Farooq S, Mehmood T, Reyes M, Samadani U. Actual and projected incidence rates for chronic subdural hematomas in United States Veterans Administration and civilian populations. J Neurosurg. 2015 Nov;123(5):1209-15. doi: 10.3171/2014.9.JNS141550. Epub 2015 Mar 20. PMID 25794342
- [Background] Baechli H, Nordmann A, Bucher HC, Gratzl O. Demographics and prevalent risk factors of chronic subdural haematoma: results of a large single-center cohort study. Neurosurg Rev. 2004 Oct;27(4):263-6. doi: 10.1007/s10143-004-0337-6. Epub 2004 May 18. PMID 15148652
- [Background] Yang S, Zhang X, Jin Y. Spontaneous resolution of nontraumatic chronic subdural hematoma associated with anti-aggregation therapy. J Craniofac Surg. 2014 Jul;25(4):e363-5. doi: 10.1097/SCS.0000000000000814. PMID 25006949
- [Background] Berghauser Pont LM, Dippel DW, Verweij BH, Dirven CM, Dammers R. Ambivalence among neurologists and neurosurgeons on the treatment of chronic subdural hematoma: a national survey. Acta Neurol Belg. 2013 Mar;113(1):55-9. doi: 10.1007/s13760-012-0130-1. Epub 2012 Sep 14. PMID 22975837
- [Background] Brennan PM, Kolias AG, Joannides AJ, Shapey J, Marcus HJ, Gregson BA, Grover PJ, Hutchinson PJ, Coulter IC; British Neurosurgical Trainee Research Collaborative. The management and outcome for patients with chronic subdural hematoma: a prospective, multicenter, observational cohort study in the United Kingdom. J Neurosurg. 2017 Oct;127(4):732-739. doi: 10.3171/2016.8.JNS16134. Epub 2016 Nov 11. PMID 27834599
- [Background] Forster MT, Mathe AK, Senft C, Scharrer I, Seifert V, Gerlach R. The influence of preoperative anticoagulation on outcome and quality of life after surgical treatment of chronic subdural hematoma. J Clin Neurosci. 2010 Aug;17(8):975-9. doi: 10.1016/j.jocn.2009.11.023. Epub 2010 May 23. PMID 20580997
- [Background] Bacigaluppi S, Guastalli F, Bragazzi NL, Balestrino A, Bruzzi P, Zona G. Prognostic factors in chronic subdural hematoma: results from a monocentric consecutive surgical series of 605 patients. J Neurosurg Sci. 2021 Feb;65(1):14-23. doi: 10.23736/S0390-5616.17.04103-0. Epub 2017 Sep 28. PMID 28959873
- [Background] Poulsen FR, Munthe S, Soe M, Halle B. Perindopril and residual chronic subdural hematoma volumes six weeks after burr hole surgery: a randomized trial. Clin Neurol Neurosurg. 2014 Aug;123:4-8. doi: 10.1016/j.clineuro.2014.05.003. Epub 2014 May 14. PMID 25012003
- [Background] Berghauser Pont LM, Dirven CM, Dippel DW, Verweij BH, Dammers R. The role of corticosteroids in the management of chronic subdural hematoma: a systematic review. Eur J Neurol. 2012 Nov;19(11):1397-403. doi: 10.1111/j.1468-1331.2012.03768.x. Epub 2012 May 29. PMID 22642223
- [Background] Stary JM, Hutchins L, Vega RA. Tranexamic Acid for Recurring Subdural Hematomas Following Surgical Evacuation: A Clinical Case Series. J Neurol Surg A Cent Eur Neurosurg. 2016 Sep;77(5):422-6. doi: 10.1055/s-0036-1584212. Epub 2016 Jun 14. PMID 27300772
- [Background] Kageyama H, Toyooka T, Tsuzuki N, Oka K. Nonsurgical treatment of chronic subdural hematoma with tranexamic acid. J Neurosurg. 2013 Aug;119(2):332-7. doi: 10.3171/2013.3.JNS122162. Epub 2013 May 3. PMID 23641825
- [Background] Tanweer O, Frisoli FA, Bravate C, Harrison G, Pacione D, Kondziolka D, Huang PP. Tranexamic Acid for Treatment of Residual Subdural Hematoma After Bedside Twist-Drill Evacuation. World Neurosurg. 2016 Jul;91:29-33. doi: 10.1016/j.wneu.2016.03.062. Epub 2016 Mar 29. PMID 27032521
- [Background] Kutty RK, Peethambaran AK, Sunilkumar, Anilkumar M. Conservative Treatment of Chronic Subdural Hematoma in HIV-Associated Thrombocytopenia with Tranexamic Acid. J Int Assoc Provid AIDS Care. 2017 May/Jun;16(3):211-214. doi: 10.1177/2325957416680294. Epub 2016 Dec 1. PMID 27909114
- [Background] Wakabayashi Y, Yamashita M, Asano T, Yamada A, Kenai H, Kondoh Y, Hori Y, Nagatomi H. [Effect of Gorei-san with tranexamic acid for preventing recurrence of chronic subdural hematoma]. No Shinkei Geka. 2012 Nov;40(11):967-71. Japanese. PMID 23100384
- [Background] Iorio-Morin C, Blanchard J, Richer M, Mathieu D. Tranexamic Acid in Chronic Subdural Hematomas (TRACS): study protocol for a randomized controlled trial. Trials. 2016 May 5;17(1):235. doi: 10.1186/s13063-016-1358-5. PMID 27150916
- [Background] Germans MR, Post R, Coert BA, Rinkel GJ, Vandertop WP, Verbaan D. Ultra-early tranexamic acid after subarachnoid hemorrhage (ULTRA): study protocol for a randomized controlled trial. Trials. 2013 May 16;14:143. doi: 10.1186/1745-6215-14-143. PMID 23680226
- [Background] Parker RI, Hagan-Burke S. Useful effect size interpretations for single case research. Behav Ther. 2007 Mar;38(1):95-105. doi: 10.1016/j.beth.2006.05.002. Epub 2006 Dec 8. PMID 17292698
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Myles PS, Smith JA, Forbes A, Silbert B, Jayarajah M, Painter T, Cooper DJ, Marasco S, McNeil J, Bussieres JS, McGuinness S, Byrne K, Chan MT, Landoni G, Wallace S; ATACAS Investigators of the ANZCA Clinical Trials Network. Tranexamic Acid in Patients Undergoing Coronary-Artery Surgery. N Engl J Med. 2017 Jan 12;376(2):136-148. doi: 10.1056/NEJMoa1606424. Epub 2016 Oct 23. PMID 27774838
- [Background] Lin Z, Xiaoyi Z. Tranexamic acid-associated seizures: A meta-analysis. Seizure. 2016 Mar;36:70-73. doi: 10.1016/j.seizure.2016.02.011. Epub 2016 Feb 26. PMID 26967164
- [Background] Berntorp E, Follrud C, Lethagen S. No increased risk of venous thrombosis in women taking tranexamic acid. Thromb Haemost. 2001 Aug;86(2):714-5. No abstract available. PMID 11522029
- [Background] Gaillard S, Dupuis-Girod S, Boutitie F, Riviere S, Moriniere S, Hatron PY, Manfredi G, Kaminsky P, Capitaine AL, Roy P, Gueyffier F, Plauchu H; ATERO Study Group. Tranexamic acid for epistaxis in hereditary hemorrhagic telangiectasia patients: a European cross-over controlled trial in a rare disease. J Thromb Haemost. 2014 Sep;12(9):1494-502. doi: 10.1111/jth.12654. Epub 2014 Jul 29. PMID 25040799
- [Background] M Versteegh M, M Vermeulen K, M A A Evers S, de Wit GA, Prenger R, A Stolk E. Dutch Tariff for the Five-Level Version of EQ-5D. Value Health. 2016 Jun;19(4):343-52. doi: 10.1016/j.jval.2016.01.003. Epub 2016 Mar 30. PMID 27325326
- [Derived] Immenga S, Lodewijkx R, Roos YBWEM, Middeldorp S, Majoie CBLM, Willems HC, Vandertop WP, Verbaan D. Tranexamic acid to prevent operation in chronic subdural haematoma (TORCH): study protocol for a randomised placebo-controlled clinical trial. Trials. 2022 Jan 18;23(1):56. doi: 10.1186/s13063-021-05907-0. PMID 35042560
- See also: cost of medicine — http://www.medicijnkosten.nl
- See also: Institute for Medical Technology Assessment — http://www.imta.nl
- See also: Central Committee on Research Involving Human Subjects (CCMO) legal frameworks, codes of conduct — https://english.ccmo.nl/investigators/legal-framework-for-medical-scientific-research/codes-of-conduct/code-of-conduct-for-health-research